CLINICAL TRIAL: NCT06855615
Title: Comparison of Thrice-Daily Premixed Human Insulin with Basal-Bolus Therapy Among Patients with Poorly Controlled Type 2 Diabetes Mellitus: a Randomised Cross-Over Study
Brief Title: Comparison of Thrice-Daily Premixed Human Insulin with Basal-Bolus Therapy Among Patients with Poorly Controlled Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Sultanah Aminah Johor Bahru (Other Government)
Collaborators: Penang Hospital, Malaysia (Other Government)
Responsible Party: Principal Investigator, Jamie Teoh Hong Im, Principal Investigator, Hospital Sultanah Aminah Johor Bahru
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-20-599-54337
Record Dates: First submitted 2025-02-17; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 Diabetes Mellitus; thrice-daily premixed human insulin (TDS PHI); basal-bolus regimen; twice-daily premixed human insulin (BD PHI); intensification therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Mixtard® 30) (Active Comparator): Participants start on TDS PHI (Mixtard® 30 TDS) and cross over to BB regimen (Insulatard® once daily plus thrice daily prandial Actrapid®) at 12 weeks (visit 4). The initial TDD of insulin equals the baseline TDD of the participants' original insulin regimen and is distributed in a 40:20:40 ratio (breakfast, lunch, and dinner).
  Interventions: Drug: Mixtard® 30 TDS; Drug: Insulatard® once daily and thrice daily prandial Actrapid®
- Group B (Insulatard® and Actrapid®) (Active Comparator): Participants start on BB regimen (Insulatard® once daily plus thrice daily prandial Actrapid®) and cross over to TDS PHI (Mixtard® 30 TDS) at 12 weeks (visit 4). The initial TDD of insulin equals the baseline TDD of the participants' original insulin regimen and is split between Actrapid® and Insulatard® as 50 and 50 per cent, respectively. Actrapid® is further divided equally across the meals.
  Interventions: Drug: Mixtard® 30 TDS; Drug: Insulatard® once daily and thrice daily prandial Actrapid®

INTERVENTIONS:
Drug: Mixtard® 30 TDS — The clinical use of TDS premixed human insulin (PHI) is unclear. In contrast, biphasic insulin analogue given thrice daily is a well-proven, safe and suitable alternative to an intensified insulin regimen.
Drug: Insulatard® once daily and thrice daily prandial Actrapid® — Basal bolus regimen is considered a physiological form of treatment and the standard of care in clinical practice but the multiple daily injections often lead to poor compliance.

SUMMARY:
The goal of this cross-over study is to learn if thrice-daily (TDS) premixed human insulin (PHI) is as useful as basal-bolus (BB) therapy as an intensification treatment in people with poorly controlled type 2 diabetes mellitus (T2DM). The main questions it aims to answer are:

* To determine the efficacy of TDS PHI compared to BB insulin regimen by measuring HbA1c changes over 12 weeks.
* To determine the changes in fasting plasma glucose (FPG), the total daily dose (TDD) of insulin, weight changes, and hypoglycaemia rate, and to study the adherence rate to insulin injection between the two regimens over 12 weeks.

Researchers will compare TDS-PHI to BB regimen to see if the glycemic control, TDD of insulin, weight gain, hypoglycemia and adherence rate are the same.

Participants will:

* take TDS-PHI or BB for 12 weeks and cross over to the other regimen for another 12 weeks
* visit the clinic once every 4 weeks for checkups and tests
* keep a diary of their self-monitoring of blood glucose (SMBG), insulin doses, hypoglycaemic symptoms and blood glucose readings, and the number of times they miss insulin injections.

DETAILED DESCRIPTION:
Thrice-daily (TDS) biphasic insulin analogues are suitable alternatives for intensifying insulin therapy, but the clinical use of TDS premixed human insulin (PHI) is unclear. When people with type 2 diabetes mellitus (T2DM) require intensification of treatment, twice daily (BD) PHI is often intensified to a basal-bolus (BB) regimen, but compliance can be poor. The investigators hypothesised that TDS PHI is as efficacious as BB therapy. A cross-over study comparing TDS PHI with BB regimens among people with T2DM is conducted primarily aimed to evaluate and compare the efficacy of TDS PHI (Mixtard® 30) with the BB insulin regimen (Insulatard® once daily plus thrice daily prandial Actrapid®) in T2DM with inadequate glycaemic control on BD PHI and to assess the changes in FPG, TDD of insulin, weight changes, hypoglycaemia rate, and rate of adherence to insulin injection in local setting. Participants receive TDS-PHI or BB for 12 weeks and cross over to the other regimen for another 12 weeks. Glycated haemoglobin (HbA1c), fasting plasma glucose (FPG), the total daily dose (TDD) of insulin, weight, hypoglycaemia, and adherence to insulin injections over 12 weeks are measured.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes patients
* Age 18 to 65 years
* HbA1c 8 to 12%
* Taking twice-daily (BD) premixed human insulin for at least 6 months

Exclusion Criteria:

* Age more than 65 years
* Had more than one episode of severe hypoglycaemia within six months
* Received treatment with systemic glucocorticoid therapy or glucose-lowering drugs other than metformin, DPP4 inhibitor and SGLT-2 inhibitor within the last three months
* Cardiac disease with a class III or class IV functional capacity
* Decompensated heart failure, unstable angina or myocardial infarction within the previous six months
* Renal insufficiency with serum creatinine more than 150umol/L
* Active liver disease or deranged liver function tests
* Untreated proliferative retinopathy or maculopathy
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of TDS PHI compared to BB insulin regimen as assessed by changes in HbA1c measured in percentage | 12 weeks

SECONDARY OUTCOMES:
Changes in FPG measured in mmol/l | 12 weeks
Changes in TDD of insulin measured in units | 12 weeks
Changes in weight measured in kilograms | 12 weeks
Changes in hypoglycemia rate as assessed by episodes per subject year | 12 weeks
Adherence to insulin injection as assessed by the frequency of missed doses per month | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamie HI Teoh, MD, Principal Investigator — Hospital Pulau Pinang, Malaysis
Locations (1):
- Hospital Pulau Pinang, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanmugasundar G, Bhansali A, Walia R, Dutta P, Upreti V. Comparison of thrice daily biphasic human insulin (30/70) versus basal detemir & bolus aspart in patients with poorly controlled type 2 diabetes mellitus - a pilot study. Indian J Med Res. 2012;135(1):78-83. doi: 10.4103/0971-5916.93428. PMID 22382187